CLINICAL TRIAL: NCT05661552
Title: Effect of Early Initiation of Evolocumab and Combination Lipid-lowering Agent on Lipid Profiles Changes in Patients With Acute Coronary Syndrome Undergoing percuTAneous coronaRy Intervention: a Prospective, Randomized Controlled Trial
Brief Title: Effect of Early Initiation of Evolocumab on Lipid Profiles Changes in Patients With ACS Undergoing PCI
Acronym: C-STAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Yongcheol Kim, Clinical Associate Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9-2022-0119
Record Dates: First submitted 2022-12-05; First posted 2022-12-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Low-Density-Lipoprotein-Type [LDL] Hyperlipoproteinemia
Keywords: acute coronary syndrome; low-density-lipoprotein; PCSK9 inhibitor
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — evolocumab; Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Intervention Model Description: The experimental and control groups consist of patients undergoing stenting for acute coronary syndrome and will be randomized to receive early evolocumab along with statin/ezetimibe use or no evolocumab. Rosuvastatin 5 mg and Ezetimibe 10 mg are administered to both the experimental group and the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab treatment group (Experimental): The experimental group will receive Rosuvastatin 5 mg, Ezetimibe 10 mg, and evolocumab by subcutaneous injection. Evolocuumab will be administered at a dose of 140 mg once during the study period.
  Interventions: Drug: Evolocumab 140 MG/ML; Drug: Rosuvastatin 5mg; Drug: Ezetimibe 10mg
- Group not receiving evolocumab (Active Comparator): The control group receives Rosuvastatin 5 mg and Ezetimibe 10 mg.
  Interventions: Drug: Rosuvastatin 5mg; Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Evolocumab 140 MG/ML — Randomly assigned Evolocumab + rosuvastatin + ezetimibe versus rosuvastatin + ezetimibe
  Other Names: REPATHA® (Amgen Inc, Thousand Oaks, California, USA)
  Arms: Evolocumab treatment group
Drug: Rosuvastatin 5mg — Rosuvastatin 5mg will be assigned to all participants
Drug: Ezetimibe 10mg — Ezetimibe 10mg will be assigned to all participants

SUMMARY:
Investigators aimed to evaluate efficacy and safety of early Initiation of evolocumab and combination lipid-lowering agent (statin + Ezetimibe) on lipid profiles changes in patients with ACS undergoing PCI

DETAILED DESCRIPTION:
Recently, studies have reported that strong LDL cholesterol lowering through PCSK9 inhibitors early in patients with acute myocardial infarction under coronary intervention results in plaque stability as well as plaque regression, which is the cause of arteriosclerosis in the coronary artery. However, the LDL cholesterol reduction effect on statin is different from that of Westerners and Asians, and studies on the LDL cholesterol reduction effect of Koreans on the early use of PCSK9 inhibitors are insufficient. Therefore, we would like to study the effect of reducing LDL cholesterol by administering Evolocumab early after the procedure in patients who underwent percutaneous coronary stent insertion for acute coronary syndrome in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Over 19 years old
2. Patients who agreed to the research protocol and clinical follow-up survey plan, decided to participate in this study voluntarily, and gave written consent to the informed consent form.
3. Patients who underwent percutaneous coronary stenting for acute coronary syndrome

Exclusion Criteria:

1. Patients who have previously taken statins,
2. Patients with active liver disease or patients with three times or more increase in AST or ALT
3. If you have an allergic or hypersensitivity reaction to Evorucumab, statin, or Ezetimib,
4. Pregnant women, lactating women, or women of childbearing age who plan to become pregnant during this study
5. The remaining life expectancy is expected to be less than a year.
6. Subjects who visited the hospital due to psychogenic shock and are expected to be less likely to survive by medical judgment
7. Subjects participating in a randomized clinical trial of medical devices/pharmaceuticals

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL level (%) | Baseline, 2 weeks later
  Difference in LDL level change between baseline and 2 weeks later in the test group and control group

SECONDARY OUTCOMES:
Percent change in LDL level (%) | baseline, 2 weeks later 4 weeks later
  Percent change in LDL level 2 weeks and 4 weeks later compared to baseline in the test group and control group
Differences in LDL level change (mg/dL) | baseline, 2 weeks later 4 weeks later
  Differences in LDL level change compared to Baseline between test and control groups
Presence or absence of side effects | baseline, 2 weeks later 4 weeks later
  Presence or absence of side effects (muscle pain, digestive disturbance, test abnormalities) after 2 weeks and 4 weeks of discharge compared to baseline in the test group and control group
Liver function test including Aspartate aminotransferase(AST)/alanine aminotransferase(ALT) (IU/L) level | baseline, 2 weeks later 4 weeks later
  Liver function test including Aspartate aminotransferase(AST)/alanine
Creatine kinase(CK) (IU/L) | baseline, 2 weeks later 4 weeks later
  Creatine kinase(CK) (IU/L)
C-Reactive Protein(CRP) (mg/L) | baseline, 2 weeks later 4 weeks later
  C-Reactive Protein(CRP) (mg/L)
Lipoprotein(a) (nmol/L) | baseline, 2 weeks later
  Lipoprotein(a) (nmol/L)
HbA1c(%) level | baseline, 4 weeks later
  HbA1c level at 4 weeks later compared to baseline in the test group and control group
Cognitive function analysis | 2 weeks later
  Patients perform self-assessment using a 23-item questionnaire that represents the execution and memory area subscales of all short-lived recognition (ECOG) tools. The cognitive functional analysis scale is evaluated on a 5-point scale, and the lower the score, the better the functional scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yongcheol Kim, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roh JW, Lee OH, Kim Y, Heo SJ, Im E, Cho DK. Effect of Early Initiation of Evolocumab on Lipid Profiles Changes in Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention. Korean Circ J. 2026 Jan 6. doi: 10.4070/kcj.2025.0315. Online ahead of print. PMID 41560483